CLINICAL TRIAL: NCT06699862
Title: The Use of Competition to Increase the Engagement in a Time-efficient School-based Intervention for Increasing Cardiorespiratory Fitness in Older Adolescents: the Burn 2 Learn - Mallorca Cluster Randomized Controlled Trial
Brief Title: The Use of Competition in a School-based Intervention for Increasing Cardiorespiratory Fitness in Adolescents
Acronym: B2L-M
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 385CER23
Record Dates: First submitted 2024-11-07; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cardiorespratory Fitness; Mental Health; School-based Intervention
MeSH Terms: conditions — Psychological Well-Being | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): During the 10-week intervention period, the control group will continue their regular physical education (PE) classes, taught by the schools' PE teachers following the standard curriculum.
- Experimental condition 1: HIIT without competition (HIIT) (Experimental): In the experimental group, Burn 2 Learn - Mallorca (B2L-M) HIIT sessions will be incorporated into regular PE classes twice a week, delivered by the schools' PE teachers. Each session will last 8-10 minutes at the start of class and include a brief warm-up with a mix of aerobic and bodyweight muscle-strengthening exercises. The sessions are designed to be both vigorous and enjoyable to maximize student engagement.
  Interventions: Behavioral: High Intensity Interval Training
- Experimental condition 2: HIIT with competition (HIIT+C) (Experimental): A key challenge of HIIT is motivating students to maintain high-intensity effort (≥85% of maximum heart rate). To address this, the second experimental condition introduces a competitive element as a motivational strategy. Students will participate in a 10-week school competition to earn points for their class. During each HIIT session, heart rate data will be tracked to monitor exercise intensity and calculate competition points. Each class will earn points equal to the total minutes of vigorous exercise (≥85% of maximum heart rate) achieved collectively by its members.
  The competition focuses exclusively on effort rather than physical fitness, ensuring that all participants can contribute equally regardless of their initial fitness levels. This approach emphasizes engagement and teamwork while encouraging students to give their best effort during the sessions.
  Interventions: Behavioral: High Intensity Interval Training with Competition

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Throughout the 10-weeks intervention period, B2L-M HIIT sessions will be delivered during regular PE classes twice a week, by the schools' PE teachers. The HIIT sessions will be applied in the first 8-10 min of each PE class, including a brief warm-up involving a combination of aerobic and body weight muscle-strengthening exercises, and designed to be fun and engaging as well as vigorous in nature
  Arms: Experimental condition 1: HIIT without competition (HIIT)
Behavioral: High Intensity Interval Training with Competition — Students will participate in a school competition to win points for their class for a 10-week period. In every HIIT session the heart rate will be tracked to measure the exercise intensity and also it will be used to win points for the competition. Every class will receive the same number of points as the sum of the minutes of exercise at a vigorous intensity (i.e., ≥85% max. heart rate) of each participant. This fact means that the physical fitness is irrelevant to the competition aspect, which will only consider the effort of the participants.
  Arms: Experimental condition 2: HIIT with competition (HIIT+C)

SUMMARY:
Regular physical activity offers numerous physical, psychological, and cognitive health benefits. However, physical inactivity among adolescents remains a global concern, with 81% of 11- to 17-year-olds failing to meet WHO's recommendation of at least one hour of moderate- to vigorous-intensity activity daily. This inactivity contributes to immediate and long-term health risks, as many non-communicable diseases (NCDs) in adulthood are linked to behaviors established during adolescence. Promoting healthy lifestyles early is crucial for lifelong health and disease prevention.

One significant barrier to effective school-based physical activity programs, such as High-Intensity Interval Training (HIIT), is maintaining student motivation. Low engagement often results in poor adherence. Integrating competition-focused on effort rather than performance-may enhance student participation and make HIIT interventions more effective and easier to implement.

This study will evaluate the impact of competition on the Burn 2 Learn - Mallorca (B2L-M) program, targeting adolescents aged 15-18. The intervention aims to determine whether competition improves engagement and outcomes compared to non-competitive groups. The primary outcome is cardiorespiratory fitness (CRF), while secondary outcomes include muscular strength, physical activity levels, body composition, mental health (stress and sleep quality), behavior change mediators (self-efficacy, motivation), on-task behavior, blood pressure, and sitting posture.

The B2L-M intervention will involve a 16-week, three-arm cluster randomized controlled trial in Mallorca, Spain, recruiting approximately 360 students from six schools. The program includes teacher-led HIIT sessions twice weekly during physical education, supported by information seminars, a dedicated website, and parental e-newsletters. Outcomes will be assessed at baseline and after 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Students who belong from "3º ESO" to "1º bachillerato" levels

Exclusion Criteria:

* Students with a health or medical condition that would preclude participation in vigorous physical activity will be excluded from the study but will still participate in normal lessons adapted by the PE teacher

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 10 weeks
  CRF will be assessed using the ALPHA (Assessing Levels of Physical Fitness and Health in Adolescents) health-related fitness test battery for children and adolescents. Participants are required to run between two lines 20 m apart in time with an audio signal. The initial speed of the signal is 8.5 km/h and increases by 0.5 km/h per minute. The test ends when the participant fails to reach the end lines in sync with the audio signal on two consecutive occasions or stops due to fatigue. The total number of laps will be used to estimate maximal aerobic capacity (i.e., VO₂ max).

SECONDARY OUTCOMES:
Physical activity | 10 weeks
  The investigators will assess physical activity using tri-axial ActiGraph wGT3X-BT accelerometers (ActiGraph LLC, Pensacola, FL, USA). ActiGraph sensors have been widely studied and shown adequate reproducibility, validity and feasibility for children and adolescents. Participants will wear the accelerometer for seven consecutive days, including weekdays and weekends, except during water-based activities such as swimming or showering. The device will be worn on the wrist of the non-dominant hand. This technique is one of the most reliable methods to quantitatively record and store physical activity data. Physical activity intensity will be categorized into light, moderate, and vigorous levels based on established thresholds.
Musculoskeletal fitness (muscular strength) | 10 weeks
  Lower body musculoskeletal fitness will be assessed through the standing long jump test, which is considered a general index of muscular fitness in youth. Participants will jump as far as they can from a starting point behind a marked line.
Waist circumference | 10 weeks
  Waist circumference will be measured in centimeters using a non-extendible steel tape.
Height | 10 weeks
  Height will be measured in centimeters using a portable stadiometer.
Weight | 10 weeks
  Weight will be measured in kilograms using a portable digital scale.
Body Mass Index (BMI) | 10 weeks
  Weight and height will be combined to report BMI in kg/m^2).
Chronic stress | 10 weeks
  Chronic stress levels will be analyzed in a sub-sample of students (n = 200). Stress can be accurately assessed by determining the accumulation of cortisol within the hair shaft using a sample taken from the vertex at the back of the head. As human hair grows at approximately 1 cm per month, each cm reflects the stressors experienced in the corresponding month. Cortisol concentrations will be determined from the 3 cm hair segment closest to the scalp, representing cumulative stress levels over the previous 2-3 months. The intra-individual stability (r = 0.68-0.79) and validity of hair cortisol as a retrospective measure of stress are well-supported in the adolescent literature.
Perceived stress | 10 weeks
  Perceived stress will be self-reported using the European Spanish version of the Perceived Stress Scale, which is designed to assess the degree to which situations in one's life are stressful. Participants will be required to respond to the 10-item questionnaire in relation to the previous month. Responses are scored on a 5-point scale ranging from 0 'never' to 4 'very often' and then summing across all scale items. Higher scores indicate a greater degree of subjective stress experienced by participants
Sleep quantity and quality | 10 weeks
  Sleep quantity and quality will be objectively measured using data provided by wrist-worn accelerometry. Sleep will be analyzed according to the algorithm developed by Sadeh. Sleep quality will be represented by sleep efficiency (SE), sleep onset latency (SOL), and time awake per hour after sleep onset (TAPH).
Self-reported sleep quality | 10 weeks
  The Spanish version of the self-reported Pittsburgh Sleep Quality Index (PSQI) will be administered. This standardized clinical instrument covers a broad range of sleep quality indicators. It comprises 19 items evaluating seven components: sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and the use of sleep medication. Using a predefined formula, the PSQI score will range from 0 to 21, with higher scores indicating poorer sleep quality.
Autonomous motivation for exercise | 10 weeks
  Intrinsic (e.g., "I exercise because it's fun") and identified (e.g., "I value the benefits of exercise") motivation will be assessed using subscales from the Spanish version of the Behavioral Regulations in Exercise Questionnaire. Responses will be scored on a 5-point scale ranging from 0, "Not true for me," to 4, "Very true for me."
On-task behaviour | 10 weeks
  On-task and off-task behavior will be assessed during regular classroom activities using established observation methods. Trained research assistants will conduct 30-minute classroom observations (starting 5 minutes after students enter). They will assess six randomly selected students per session (5 minutes per student). Observers will record student behavior every 10 seconds using an observation sheet, switching to the next student after 15 seconds, and repeating this process until all students have been observed 20 times. Teachers and students will remain unaware of which students are being observed.
  On-task behavior includes actively engaging in academic tasks, such as reading, writing, or completing assigned work, as well as passively listening to teachers or peers. Off-task behavior includes motor (e.g., walking around), verbal (e.g., unrelated discussions), and passive (e.g., staring into space) actions unrelated to the task.
Blood pressure | 10 weeks
  Systolic and diastolic blood pressure will be measured using an Omron M3 Blood Pressure Monitor with a cuff size appropriate for each participant's upper arm circumference. Participants will sit quietly for 5 minutes, after which three measurements will be taken at 5-minute intervals. The analysis will use the average of the three readings.
Sitting posture | 10 weeks
  Posture will be assessed using the UPRIGHT Go Posture Training Device (Upright Technologies Ltd., Yehud, Israel). The device will be positioned at the cervicothoracic junction, just below the first prominent spinous process, using the Upright Necklace. It will record posture during an entire classroom session, reporting the percentage of time spent upright versus slouched. The device pairs with a smartphone app, enabling progress tracking toward improved posture.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain